CLINICAL TRIAL: NCT05104983
Title: Stopping TSC Onset and Progression 2B: Sirolimus TSC Epilepsy Prevention Study
Acronym: TSC-STEPS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Darcy Krueger (Other)
Responsible Party: Sponsor-Investigator, Darcy Krueger, IND Sponsor/Lead Principal Investigator, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-0438; 1R01FD007275 (FDA)
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Tuberous Sclerosis Complex; Epilepsy
Keywords: Tuberous Sclerosis Complex; TSC; epilepsy; prevention; mTOR; sirolimus; infant
MeSH Terms: conditions — Tuberous Sclerosis; Epilepsy | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: This trial will employ a randomized, double-blind, placebo-controlled multisite design to evaluate the safety and efficacy of early sirolimus treatment to prevent or delay seizure onset in TSC infants.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sirolimus (Experimental): Sirolimus
  Interventions: Drug: Sirolimus
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sirolimus — The investigational drug product to be used in this study is sirolimus, provided in oral suspension.
  Arms: Sirolimus
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This trial is a Phase II randomized, double-blind, placebo controlled multi-site study to evaluate the safety and efficacy of early sirolimus to prevent or delay seizure onset in TSC infants.

This study is supported by research funding from the Office of Orphan Products Division (OOPD) of the US Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
Tuberous Sclerosis Complex (TSC) is caused by genetic mutation in TSC1 or TSC2, resulting in dysregulation of the mechanistic target of rapamycin (mTOR) signaling pathway. Age at time of seizure onset in TSC infants has been linked to long-term neurodevelopmental outcome in this high-risk population. Sirolimus is an mTOR inhibitor used to treat many of the symptoms of TSC, including epilepsy. This will be the first study to truly evaluate a targeted, disease-modifying drug therapy for preventing or delaying seizure onset in TSC using a rational, mechanism-based therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

1. 0-6 months of age at the time of enrollment (subject must be <7 months of chronological age at time of randomization and treatment initiation). Corrected age must be at least 39 weeks (calculated by subtracting the number of weeks born before 40 weeks gestation from the chronological age).
2. Has a confirmed diagnosis of TSC based on established clinical or genetic criteria

Exclusion Criteria:

1. Prior history of seizures (clinical or electrographic) at the time of enrollment or identified on baseline EEG.
2. Has been treated in the past or is currently being treated at the time of enrollment with conventional anticonvulsant medications (AEDs), systemic (oral) mTOR inhibitors (such as rapamycin, sirolimus, or everolimus), ketogenic-related special diet, or another anti-seizure therapeutic agent, device, or procedure.
3. Has taken any other investigational drug as part of another research study, within 30 days prior to the baseline screening visit.
4. Has a significant illness or active infection at the time of the baseline screening visit
5. Has a history of significant prematurity, defined as gestational age <30 weeks at the time of delivery, or other significant medical complications at birth or during the neonatal period that other than TSC would convey additional risk of seizures or neurodevelopmental delay (i.e. HIE, severe neonatal infection, major surgery, prolonged ventilatory or other life-saving supportive care or procedures).
6. Abnormal laboratory values at baseline (i.e., renal function, liver function, or bone marrow production) that are in the opinion of the investigator clinically significant and may jeopardize the safety of the study subject.
7. Prior, planned or anticipated neurosurgery within 3 months of the baseline visit
8. Has a TSC-associated condition for which mTOR treatment is clinically indicated (i.e. SEGA or AML).
9. Subjects who are, in the opinion of the investigator, unable to comply with the requirements of the study.

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy -- time to seizure onset | 12 months of age
  Time to seizure onset, comparing sirolimus with placebo
Safety -- adverse events | 12 months of age
  Percentage of subjects reporting severe (CTCAE v5.0 grade >= 3) adverse event (AE) or serious adverse event (SAE), comparing sirolimus with placebo.

SECONDARY OUTCOMES:
Neurodevelopmental Outcomes | 12 and 24 months of age
  Neurodevelopmental outcomes at the end of treatment, comparing sirolimus with placebo.
Quality of Life Outcomes | 12 and 24 months of age
  Patient and caregiver quality of life, comparing sirolimus with placebo.
EEG Biomarkers | 12 and 24 months of age
  EEG measures of neuronal connectivity, comparing sirolimus with placebo.
MRI Biomarkers | 12 and 24 months of age
  MRI measures of neuronal connectivity, comparing sirolimus with placebo.
Sirolimus Precision Dosing | 12 months of age
  Validate the feasibility and effectiveness of sirolimus precision dosing in infants with TSC

CONTACTS AND LOCATIONS:
Overall Officials: Darcy A Krueger, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Martina Bebin, MD, MPA, Principal Investigator — University of Alabama at Birmingham
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University -- St. Louis, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Texas HSC at Houston, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington